CLINICAL TRIAL: NCT03572309
Title: Incidence of Trauma Induced Coagulopathy in Patients With Prehospital Administration of Fibrinogen
Acronym: TICAF
Status: Completed | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CT0022018
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Trauma; Hemorrhage; Coagulopathy
Keywords: trauma induced coagulopathy; multiple trauma; fibrinogen
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Hemostatic Disorders; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the study is to find out the incidence of trauma induced coagulopathy in patients with severe trauma who received fibrinogen prior admission to emergency department during prehospital care.

DETAILED DESCRIPTION:
The study will commence following the Approval by The Ethics Research Committee. All patients admitted to emergency department during the study will be enrolled after fulfilling the inclusion criteria and in the absence of any exclusion criteria. Informed consent will be requested. After admission to emergency department the blood samples will be taken and blood tests and viscoelastic tests will be performed. All data and results will be entered in the study form. Statistical analysis will be performed and incidence of trauma induced coagulopathy estimated. In addition, 28-day mortality and the incidence of thromboembolic complications will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* multiple trauma, injury severity score (ISS) ≥16
* administration of fibrinogen in prehospital care
* age 18-80 years

Exclusion Criteria:

* ISS 75
* pregnancy
* therapeutic anticoagulation
* therapeutic antiaggregation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult trauma patients with severe trauma admitted to emergency departement of university hospital who recieved fibrinogen during prehospital care.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Trauma induced coagulopathy | day of enrolment
  Incidence of trauma induced coagulopathy

SECONDARY OUTCOMES:
28day mortality | 28 days after enrolment
thromboembolic complications | 28 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, MD, PhD, Study Chair — Masaryk University
Locations (1):
- University Hospital Brno and Masaryk University Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No